CLINICAL TRIAL: NCT06596044
Title: Suicide Prevention In Department of Veterans Affairs Community Care Network Mental Health Settings
Brief Title: Suicide Prevention After Community Care Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MHBC-003-24S; 101CX002797 (Other Grant/Funding Number: VA Office of Research and Development)
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Suicide Prevention
Keywords: Mental health education; Clinical trial; Suicidal ideation; Suicide, attempted; Self-injurious Behavior; Suicide; Suicide Prevention
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation; Suicide, Attempted; Self-Injurious Behavior; Suicide | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel: VA BIC plus standard care vs. standard care alone
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to treatment allocation and will remind the participant at each contact to not disclose their treatment status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VA BIC (Experimental): Patients randomized to VA BIC will receive the VA BIC intervention plus standard care
  Interventions: Behavioral: VA BIC; Other: Standard Care
- Standard Care (Other): Patients randomized to the control arm will receive standard care alone.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: VA BIC — VA BIC is a suicide prevention strategy that is designed to meet the needs of Veterans who receive acute psychiatric treatment. VA BIC can be delivered by a trained mental health provider (e.g., mental health nurse, social worker, psychologist, psychiatrist). VA BIC includes two synergistic elements to support the patient after a mental health discharge. The elements include a brief educational session, where the patient receives a one-on-one, one-hour, personalized educational session on suicide prevention. The session incorporates aspects of motivational interviewing. The patient then receives 7 regular follow-up contacts that are conducted by the interventionist. Here the interventionist monitors symptoms, assesses treatment adherence, reviews the safety plan, and assists the patient with engaging in steps to promote their well-being. The sessions incorporate aspects of motivational interviewing. Of note patients in this arm will also receive standard care.
  Arms: VA BIC
Other: Standard Care — Regardless of study assignment, all patients will have access to standard care provided upon mental health discharge in non-VA settings. VA staff will also follow standard procedures for mitigating risk including placing Veterans on high risk list when clinically appropriate.

SUMMARY:
The study is of high importance to Veterans' health because it will study a suicide prevention intervention in a Veteran population that is at high risk of suicide but has not been a specific focus of the Veteran Affairs' (VA's) suicide prevention efforts. Specifically, a growing number of Veterans are now receiving acute mental health treatment in VA-purchased settings (commonly referred to as Community Care). While these Veterans are at high risk of suicide after discharge, very little is known about how to prevent suicide in these Veterans. This study will directly address this problem by looking at whether a promising suicide prevention strategy called the VA Brief Intervention and Contact Program (VA BIC) can decrease the risk of suicide in Veterans after they are discharged from a non-VA mental health treatment setting. The proposed research is highly pertinent to the VA's top clinical priority-to prevent suicide in Veterans.

DETAILED DESCRIPTION:
Background: Suicide is a chief concern in Veterans. An increasing number of Veterans are accessing acute psychiatric treatment in non-VA settings. There is little knowledge about effective strategies to mitigate suicide risk in this population. A promising suicide prevention strategy, called the VA Brief Intervention and Contact Program (BIC), has been developed. VA BIC is designed to meet the unique needs of Veterans. Pilot studies of VA BIC in VA settings have suggested that VA BIC may address key factors related to suicide risk during care transitions including social connectedness and treatment engagement. Based on these promising results and given the critical gaps in suicide prevention care in Veterans who receive acute psychiatric treatment in non-VA settings, it is essential to determine whether VA BIC can reduce suicide risk in this high-risk population.

Objectives: This project aims to 1) Identify the effect of VA BIC on suicidal ideation after a non-VA mental health discharge, compared to standard care alone; 2) Identify the effect of VA BIC on engagement in mental health care after a non-VA mental health discharge, compared to standard care alone; 3) Identify the effect of VA BIC on social connectedness after a non-VA mental health discharge, compared to standard care alone; and 4) Compare the effect of VA BIC on suicidal behavior after a non-VA mental health discharge, compared to standard care alone.

Methods: This is an assessor-blinded, randomized control trial of VA BIC plus standard care compared to standard care alone. The trial will enroll up to 120 participants aged 18 years and older who are Veterans eligible to receive VA services and have received acute psychiatric treatment in non-VA settings affiliated with VA in Northern New England. Participants will be randomized to either the VA BIC intervention plus standard care or standard care alone. Suicidal ideation, engagement in mental health care, social connectedness and suicidal behavior will be measured at baseline and three, six , and nine months follow-up.

Hypothesis: Veterans receiving the VA BIC intervention plus standard care will report reductions in suicidal thoughts at follow-up assessments compared to Veterans receiving standard care alone. Veterans receiving the VA BIC intervention plus standard care will experience an increase in engagement in mental health care and social connectedness at follow-up assessments compared to Veterans receiving standard care alone

ELIGIBILITY:
Inclusion Criteria:

* Veteran who is eligible to receive VA services;
* 18 years or older;
* able to speak English;
* received acute psychiatric treatment in a non-VA setting affiliated with VA in Northern New England;
* endorse recent suicidal ideation (score 2+ on Beck Scale for Suicidal Ideation).

Exclusion Criteria:

* Unable to provide informed consent;
* Currently receiving assertive community treatment;
* Potentially vulnerable populations including prisoners, institutionalized patients, or patients currently admitted on involuntary commitment status;
* Study physician deems the patient is not clinically appropriate because of clinical status such as presence of active psychosis or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation: The Beck Scale for Suicidal Ideation (BSS) | Baseline to 9 months post-baseline
  The Beck Scale for Suicidal Ideation (BSS) is a self-reported, 21-item scale that assesses symptoms of suicidal ideation. The total score ranges from 0-38. While there is no established BSS cutoff score to classify suicide risk, there is evidence that higher scores on the BSS correspond to more severe suicidal ideation and that a change of five points or more on the total BSS scores may be clinically relevant.

SECONDARY OUTCOMES:
Mental Healthcare Utilization: The number of mental health visits attended | Baseline to 3 months post-baseline
  The investigators will measure the total number of mental health visits that patients attended. The investigators will abstract these data from the electronic medical record. Because some patients may attend mental health visits outside of the VA healthcare system, the investigators will use a standardized data collection form to ask patients to self-report on any non-VA mental health visits they attended.
Patient perception of ability to cope with suicidal behavior: The Suicide-Related Coping Scale (SRCS) | Baseline to 9 months post-baseline
  The Suicide-Related Coping Scale (SRCS) is a self-reported, 17-item scale that assesses a patient's perception of their ability to manage suicidal behavior. The scale includes two-subscales including an External Coping subscale (7-items) and an Internal Coping subscale (7-items). The total scores on the SRCS range from 0-68. The total scores on the subscales range from 0-28 for the External Coping subscale and 0-28 for the Internal Coping subscale. Higher scores indicate greater belief in ability to cope with suicidal behavior.
Social Connectedness: Interpersonal Needs Questionnaire-15 (INQ-15) | Baseline to 9 months post-baseline
  The Interpersonal Needs Questionnaire-15 (INQ-15) is a self-reported, 15-item scale that assesses a patient's perception of their connectedness with others. The total scores range from 15- 105. The scale includes two-subscales: a Thwarted Belongingness subscale (9-items) and a Perceived Burdensomeness subscale (6-items) that are used to assess different aspects of connectedness. The total scores on the Thwarted Belongingness subscale range from 9-63. The total scores on the Perceived Burdensomeness subscale range from 6-42. Higher scores indicate worse perceived connectedness.
Suicide Attempt Events: Fatal and non-Fatal Suicide Attempts | Baseline to 9 months post-baseline
  The investigators will measure the number of fatal and non-fatal suicide attempts. The investigators will report the number of patients who experience at least one suicide attempt (fatal and non-fatal). To assess for suicide attempts (fatal/non-fatal), the investigators will use the subpart of the Columbia Suicide Severity Rating Questionnaire (C-SSRS). This is a valid measure of suicidal behavior. The investigators will also review the medical record for reports of suicide attempts (fatal/non-fatal). Of note the subpart of the C-SSRS that assesses for suicidal behavior including suicide attempts does not generate a score. It only reports on the occurrence of the event.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Riblet, MD MPH, Principal Investigator — White River Junction VA Medical Center, White River Junction, VT
Locations (1):
- White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont, United States

IPD SHARING:
Plan to Share IPD: No